CLINICAL TRIAL: NCT01412593
Title: Intra-hepatic Artery Bone Marrow Derived Stem Cells Infusion for the Treatment of Advanced Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Dr Ayman Abdo, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDRC001SC
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-05

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem cell transplant (Experimental)
  Interventions: Biological: Stem cell transplant
- Control (No Intervention)

INTERVENTIONS:
Biological: Stem cell transplant — Patients randomized to the intervention arm will be admitted to the Liver Care Unit. Granulocyte colony-stimulating factor (G-CSF; 300mcg/mL) will be administered for 1 day as a single daily subcutaneous dose. This dose is sufficient to induce 10 folds enrichment for bone marrow cells.
  Arms: Stem cell transplant

SUMMARY:
Liver disease is a common medical problem in Saudi Arabia. Early studies indicated that around 10% of the Saudi population is either infected with hepatitis B or C. An estimated 12% of chronic HCV and HBV patients undergoing liver biopsy from Saudi centers have cirrhosis. Of these 3-5% would decompensate yearly thereby requiring liver transplantation. Based on the most recent national census figures, and a 1-2% prevalence rate of HBV and HCV nationwide, an estimated 1,000 patients would require liver transplantation on a yearly basis for decompensated cirrhosis.

Liver transplantation is the only available life saving treatment for patients with end stage liver disease. Unfortunately less than 100 liver transplantations are performed in Saudi Arabia in three centers. Around 100 other patients travel abroad for transplantation annually while all other patients progressively deteriorate and eventually die from the complications of decompensated liver cirrhosis.

In addition, even in patients who are listed for liver transplantation, often patients are too sick to wait on the transplant list that often takes more than a year and the on-list mortality is high. A procedure or an intervention that may help to stabilize liver function in order to help patients survive on the transplant list while awaiting liver transplantation would be of immense benefit. Examples of such interventions are already approved and used in some centers like the MARS system.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinically diagnosed liver cirrhosis by any of the following: ultrasound/MRI/ CT/ + tissue biopsy.
* MELD score ≥ 18 and <35
* Ability to sign an informed consent
* Refused by liver transplant program or labeled as not a liver transplant candidate, decided by at least 3 transplant physicians

Exclusion Criteria:

* On a liver transplantation waiting list
* Questionable diagnosis of cirrhosis
* Prior history of organ transplantation
* Past history of malignancy within the 2 years prior to inclusion
* Probable or diagnosis of hepatocellular carcinoma
* Major hepatic vascular thrombosis (hepatic artery, or portal or hepatic veins)
* Serious cardiovascular or respiratory disease, or other medical condition with a high anticipated mortality within twelve months
* Current or recent (within the past 4 weeks) use of vasoactive drugs (Epinephrine, Norepinephrine, Vasopressin, Dopamine, terlipressin)
* Type-1 (acute) hepatorenal syndrome
* Levels of serum creatinine >150 µmol/ml and/or creatinine clearance <30 ml/min (as calculated by MDRD system)
* Documented or suspected ongoing infection
* Active or recent gastrointestinal bleeding episode (in the previous 4 weeks)
* Active alcohol abuse extending to within the previous six months
* Pulmonary hypertension (PAP > 35 mmHg), porto-pulmonary hypertension or hepatopulmonary syndrome
* Pregnancy
* HIV infection
* Active or past drug addiction within the preceding 6 months
* History of serious or uncontrolled psychiatric disease or depression
* Contraindications to the angiography procedures (e.g. arterial aneurysm, kinking, thrombosis)
* Contraindications for bone marrow biopsy (e.g. bleeding diathesis)
* Prior shunt operative shunt procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver function measured by improvement in the model for end-stage liver disease (MELD) score. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University Hospital, Riyadh, Riyadh Region, Saudi Arabia